CLINICAL TRIAL: NCT04799353
Title: A Randomized, Double-Blind, Placebo-controlled Single-Dose Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous and Intravenous Administration of Budigalimab in Adult People Living With HIV-1 (PLWH)
Brief Title: Study to Evaluate the Safety and How the Body Handles a Single Dose of Subcutaneous (SC) and Intravenous (IV) Budigalimab in Adult Participants Living With Human Immunodeficiency Virus (HIV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-972
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus (HIV); Budigalimab; ABBV-181
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — budigalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Placebo SC + Placebo IV (Experimental): Participants will receive Subcutaneous (SC) Placebo, followed by Intravenous (IV) Placebo.
  Interventions: Drug: Placebo
- Group 2: Budigalimab (SC) + Placebo IV (Experimental): Participants will receive Subcutaneous (SC) Budigalimab, followed by Intravenous (IV) Placebo.
  Interventions: Drug: Budigalimab; Drug: Placebo
- Group 3: Budigalimab SC + Placebo IV (Experimental): Participants will receive Subcutaneous (SC) Budigalimab, followed by Intravenous (IV) Placebo.
  Interventions: Drug: Budigalimab; Drug: Placebo
- Group 4: Placebo SC + Budigalimab IV (Experimental): Participants will receive Subcutaneous (SC) Placebo, followed by IV Budigalimab.
  Interventions: Drug: Placebo; Drug: Budigalimab

INTERVENTIONS:
Drug: Budigalimab — Subcutaneous (SC)
  Other Names: ABBV-181
  Arms: Group 2: Budigalimab (SC) + Placebo IV; Group 3: Budigalimab SC + Placebo IV
Drug: Placebo — Subcutaneous (SC)
  Arms: Group 1: Placebo SC + Placebo IV; Group 4: Placebo SC + Budigalimab IV
Drug: Budigalimab — Intravenous (IV)
  Other Names: ABBV-181
  Arms: Group 4: Placebo SC + Budigalimab IV
Drug: Placebo — Intravenous (IV)
  Arms: Group 1: Placebo SC + Placebo IV; Group 2: Budigalimab (SC) + Placebo IV; Group 3: Budigalimab SC + Placebo IV

SUMMARY:
This study will evaluate how safe Budigalimab is and how it moves within the body in adult participants with HIV-1 infection.

Budigalimab is an investigational drug being evaluated for the treatment of Human Immunodeficiency Virus. Study participants will be assigned to one of the 4 treatment groups and will receive a single dose of Budigalimab or placebo subcutaneous (SC) and intravenous (IV). Around 32 participants 18-65 years of age living with Human Immunodeficiency Virus will be enrolled in the study in approximately 9 sites worldwide.

Each participant will receive single dose of SC and IV Budigalimab and/or Placebo on day 1 and will be followed for 24 weeks.

Participants will attend weekly to every two and every four weeks visits during the study at a hospital. The effect of the treatment will be checked by medical assessments, blood tests and checking for side effects. There may be higher treatment burden for participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Condition of generally good health, body mass index ≥ 18.0 to < 35.0 kg/m2.
* Laboratory values must meet acceptable criteria.
* Human Immunodeficiency Virus (HIV-1) infected on antiretroviral therapy (ART) for at least 12 months prior to screening and on current ART regimen for at least 8 weeks prior to screening.
* CD4 cell count ≥ 450 cells/μL at Screening and during the 12 months prior to Screening.
* Plasma HIV-1 RNA below the lower limit of quantification at Screening and at least 6 months prior to Screening.
* Participants agreeing to use an effective barrier method of protection (male and/or female condom) during sexual activity from Study Day 1 through last study visit for the purposes of prevention of HIV transmission.

Exclusion Criteria:

* Participants with signs/symptoms associated with SARS-CoV-2 infection OR Current SARS-CoV-2 infection by any viral nucleic acid test completed within 7 days prior to the Day 1 dose.
* Participants having history or ongoing diagnosis of acquired immunodeficiency syndrome (AIDS)-defining illness.
* Participants having history of or active immunodeficiency (other than HIV).
* Participants having active autoimmune disease or history of autoimmune disease that has required systemic treatment.
* Prior therapy/exposure to budigalimab or any other immune checkpoint inhibitor [e.g., anti-programmed cell death protein 1(PD-1), anti-PD-L1, anti-PD-L2, anti-CTLA4].
* Participants having clinically significant medical disorders that might expose the subjects to undue risk of harm, confound study outcomes, or prevent the subject from completing the study.
* Participants having active or suspected malignancy or history of malignancy (other than basal cell skin cancer or cervical carcinoma in situ) in the past 5 years.
* Participants with history of or active tuberculosis (TB) at screening.
* Participants having known psychiatric or substance abuse disorders that would interfere with adherence to study requirements.
* Participants who have received immunomodulatory or immunosuppressive (including IV/orally administered [PO] steroids at any dose, but excluding steroids that are inhaled, topical or via local injection) therapy within 24 weeks prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Study Drug-Related Grade 3 or Higher Adverse Events (AEs) | Up to approximately 24 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of the study drug as either having a reasonable possibility or no reasonable possibility. AEs are given a grade from 1-5 with Grade 3 being severe but not life-threatening and requiring hospitalization, Grade 4 being life-threatening requiring immediate intervention and Grade 5 being death related to an AE.
Number of Participants With Study Drug-Related Immune-Related Adverse Events (IRAE) | Up to approximately 24 weeks
  Assessed using the American Society of Clinical Oncology (ASCO) IRAE management guidelines [which utilizes the National Institutes of Health (NIH) Common Terminology Criteria for Adverse Events (CTCAE) grading scale] but modified, as applicable, according to the NIH Division of AIDS (DAIDS) (v2.1) AE grading scale.
Maximum Serum Concentration (Cmax) | Up to approximately 24 weeks
  Maximum Serum Concentration (Cmax) of Budigalimab.
Time to Maximum Observed Plasma Concentration (Tmax) | Up to approximately 24 weeks
  Time to Maximum Observed Plasma Concentration (Tmax) of Budigalimab.
Area Under the Plasma Concentration-time Curve (AUC) of Budigalimab in Plasma | Up to approximately 24 weeks
  Area Under the Plasma Concentration-time Curve (AUC).
Terminal Phase Elimination Half-life (t1/2) of Budigalimab in Plasma | Up to approximately 24 weeks.
  Terminal phase elimination half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (8):
  - Franco Felizarta, Md /Id# 223931, Bakersfield, California
  - Ruane Clinical Research Group /ID# 224496, Los Angeles, California
  - Quest Clinical Research /ID# 223925, San Francisco, California
  - Central Texas Clinical Research /ID# 223937, Austin, Texas
  - St. Hope Foundation, Inc. /ID# 224492, Bellaire, Texas
  - North TX Infectious Diseases /ID# 224494, Dallas, Texas
  - The Crofoot Research Center, Inc /ID# 224493, Houston, Texas
  - Peter Shalit, M.D. /ID# 224801, Seattle, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation /ID# 224230, Ponce
  - Puerto Rico AIDS Clinical Trials Unit CRS /ID# 223936, San Juan

IPD SHARING:
Plan to Share IPD: No